CLINICAL TRIAL: NCT02099253
Title: The Influence of Age on Dexmedetomidine Pharmacodynamic in Lower Extremity Surgery
Brief Title: The Influence of Age on Dexmedetomidine Pharmacodynamic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, bo xu, associate chief physician, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEX Pharmacodynamics
Record Dates: First submitted 2014-03-26; First posted 2014-03-28 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Spinal Anesthesia
Keywords: Age; Pharmacodynamics; dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Youth Group (Experimental): People in this group, aged 18~39,were accepted an initial dose of 1μg/kg, with dose adjustment intervals of 0.05μg/kg.
  Interventions: Drug: Dexmedetomidine 01
- Middle-aged Group (Experimental): People in this group, aged 40~64,were accepted an initial dose of 1μg/kg, with dose adjustment intervals of 0.05μg/kg.
  Interventions: Drug: Dexmedetomidine 01
- Older Group (Experimental): People in this group, aged 65~80,were accepted an initial dose of 0.7μg/kg, with dose adjustment intervals of 0.05μg/kg.
  Interventions: Drug: Dexmedetomidine 02

INTERVENTIONS:
Drug: Dexmedetomidine 01 — Initial doses was 1μg/kg, with dose adjustment intervals of 0.05μg/kg.
  Arms: Middle-aged Group; Youth Group
Drug: Dexmedetomidine 02 — Initial doses was 0.7μg/kg, with dose adjustment intervals of 0.05μg/kg.
  Arms: Older Group

SUMMARY:
Dexmedetomidine(DEX) is a novel , highly selective α2 adrenergic receptor agonists , and its selectivity for α2 receptor is 1600 times higher than α1.It also could provide dose-dependent sedation , analgesia , anti-anxiety and inhibition of sympathetic nerves and other effects .At earlier time It was approved by the FDA only for short-time sedation during mechanical ventilation of adult patients (<24h) in ICU. Because of its minimal impact on the respiratory , currently it was more and more widely used to sedate patients undergoing regional anesthesia.Many anesthetic pharmacokinetics and pharmacodynamics are often affected by age and gender,such as the drug sensitivity of propofol and remifentanil is increased with age,while the current study also demonstrated that gender may influence the sedate efficacy of propofol and the sensitivity of muscle loose of rocuronium. Current studies with regard to the effects of age and gender on dexmedetomidine pharmacodynamic are rare. The study is aim to explore the right DEX dose of different Age of patients to produce suitable sedation.Dexmedetomidine be used in patients with combined spinal and epidural anesthesia for sedation,which is monitored by the BIS,during the operation.The relation between BIS values and the depth of sedation for patients is also investigated.

DETAILED DESCRIPTION:
120 patients scheduled to undergo lower extremity surgery were included in one of three groups. Determination of median effective (ED50) doses was performed by the Dixon and Mood up-and-down method. Initial doses was 1μg/kg, with dose adjustment intervals of 0.05μg/kg, in the youth,and middle-aged group. The initial doses of DEX was 0.7 μg/kg,also with dose adjustment intervals of 0.05μg/kg.Sedative efficacy was defined as an OAA/S of ≤2, or an OAA/S of 3 but with an BIS value of ≤46, 26 min after the beginning of drug administration.

ELIGIBILITY:
Inclusion Criteria:

1. ASA Ⅰ ~ Ⅱ patient undergoing lower extremity surgery
2. Written informed consent from the patient or the relatives of the participating patient.
3. BMI:18.5～25

Exclusion Criteria:

1. Mental illness can not match
2. epidural anesthesia contraindicated
3. People who have Slow-type arrhythmias
4. People who were language or hearing impaired
5. Sensory block reached to T8 or higher.
6. People who had lung infection or sleep apnea syndrome.
7. Pregnancy
8. Chronic renal failure
9. Alcohol or drug abuse
10. Already taking gabapentin, pregabalin, benzodiazepin or antidepression drug

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The ED50 of DEX | 26min after the start of the infusion
  The aim of our study is to define the median effective sedative doses (ED50s) of DEX to determine the effect of age on the pharmacodynamic of DEX in lower extremity surgery using the Dixon and Mood up-and-down method。

SECONDARY OUTCOMES:
The ED95 of DEX | 26min after the start of the infusion
  To determine the optimum bolus dose (ED95) of dexmedetomidine for producing adequate sedation during spinal anesthesia in lower limb orthopedic surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Military Region General Hospital, Department of Anesthesiology, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Park SJ, Park HJ, Choi JY, Kang HS, Choi HS. The influence of age and gender on remifentanil EC(50) for preventing rocuronium induced withdrawal movements. Korean J Anesthesiol. 2010 Mar;58(3):244-8. doi: 10.4097/kjae.2010.58.3.244. Epub 2010 Mar 29. PMID 20498772
- [Background] Kodaka M, Johansen JW, Sebel PS. The influence of gender on loss of consciousness with sevoflurane or propofol. Anesth Analg. 2005 Aug;101(2):377-381. doi: 10.1213/01.ANE.0000154534.71371.4F. PMID 16037147
- [Derived] Xu B, Li Z, Zhou D, Li L, Li P, Huang H. The Influence of Age on Sensitivity to Dexmedetomidine Sedation During Spinal Anesthesia in Lower Limb Orthopedic Surgery. Anesth Analg. 2017 Dec;125(6):1907-1910. doi: 10.1213/ANE.0000000000002531. PMID 28991112